CLINICAL TRIAL: NCT06091033
Title: Perceived Stress and Black Rice (Oryza Sativa L.) Extract Fermented With Lactobacillus: a Double-blind, Randomized, Placebo-controlled Study
Brief Title: Perceived Stress and Black Rice (Oryza Sativa L.) Extract Fermented With Lactobacillus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Sang Yeoup Lee, Professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB 02-2021-041
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Perceived Stress

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fermented rice group (Experimental): This group takes black rice (Oryza Sativa L.) extract fermented with Lactobacillus for 8 weeks.
  Interventions: Dietary Supplement: Fermented rice
- Control group (Placebo Comparator): This group takes a placebo for 8 weeks.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Fermented rice — 1,000 mg of black rice (Oryza Sativa L.) extract fermented with Lactobacillus for 8 weeks
  Arms: Fermented rice group
Dietary Supplement: placebo — 1,000 mg of a placebo for 8 weeks
  Arms: Control group

SUMMARY:
The investigators will conduct a randomized, double-blind, placebo-controlled study to investigate the effects and tolerability of black rice (Oryza Sativa L.) extract fermented with Lactobacillus on patients with perceived stress for 8 weeks.

DETAILED DESCRIPTION:
A previous animal study has indicated that black rice (Oryza Sativa L.) extract fermented with Lactobacillus relieved stressful situations in a 7-week-old C57BL/6 mice model. Therefore, the investigators will conduct a randomized, double-blind, placebo-controlled study to investigate the effects and tolerability of black rice (Oryza Sativa L.) extract fermented with Lactobacillus on patients with perceived stress for 8 weeks; the safety of the compound is also evaluated. The Investigators examine stress response inventory (SRI), perceived stress scale (PSS), stress-visual analog scale (VAS), EQ-5D-5L, salivary cortisol, plasma cortisol, serotonin, dehydroepiandrosterone sulfate (DHEAS), cortisol/DHEAS ratio, adrenocorticotropic hormone (ACTH), glucose, lactate, free fatty acid (FFA), malondialdehyde (MDA) superoxide dismutase (SOD), heart rate, systolic blood pressure (BP), and diastolic BP at baseline and after 8 weeks of intervention. Eighty adults were administered either 1,000 mg of black rice (Oryza Sativa L.) extract fermented with Lactobacillus or a placebo each day for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

- the Perceived Stress Scale between 13-18

Exclusion Criteria:

* People with alcohol use/induced disorders
* Persons with brain disease or undergoing rehabilitation treatment for brain disease
* Patients with mental illnesses such as major affective disorder, post-traumatic stress disorder, uncontrolled obsessive-compulsive disorder, schizophrenia, dementia, drug addiction, etc.
* Those who have taken psychotropic drugs, sleeping pills, appetite suppressants, oral steroids, and corticosteroids within 1 month before starting the trial
* Those who have taken functional health foods recognized by the Ministry of Food and Drug Safety related to relieving tension caused by stress and improving sleep within 1 month before the start of the test
* Those who show withdrawal symptoms due to abstinence from drinking or smoking within 1 month before starting the trial.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
stress response inventory (SRI) | 8 weeks
  using SRI score. The minimum score was 0, and the maximum score was 195; higher scores mean a worse outcome.

SECONDARY OUTCOMES:
perceived stress scale (PSS) | 8 weeks
  using PSS score. The minimum score was 0, and the maximum score was 40; higher scores mean a worse outcome.
stress-Visual Analog Scale (VAS) | 8 weeks
  using stress-VAS score. The minimum score was 0, and the maximum score was 100; higher scores mean a worse outcome.
EuroQol (EQ)-5D-5L | 8 weeks
  using stress-VAS score. The minimum score was 0, and the maximum score was 1; higher scores mean a worse outcome.
Salivary cortisol (ng/dl) | 8 weeks
  Change during 8 weeks
Plasma cortisol (ng/dl) | 8 weeks
  Change during 8 weeks
Plasma serotonin (nmol/L) | 8 weeks
  Change during 8 weeks
Plasma dehydroepiandrosterone sulfate (µg/dL) | 8 weeks
  Change during 8 weeks
Plasma cortisol/dehydroepiandrosterone sulfate ratio | 8 weeks
  Change during 8 weeks
Plasma adrenocorticotropic hormone (pg/mL) | 8 weeks
  Change during 8 weeks
Fasting glucose (mg/dL) | 8 weeks
  Change during 8 weeks
Lactate (mmol/L) | 8 weeks
  Change during 8 weeks
Free fatty acid (µmol/L) | 8 weeks
  Change during 8 weeks
Heart rate (beats per minute) | 8 weeks
  Change during 8 weeks
Systolic blood pressure (BP) (mmHg) | 8 weeks
  Change during 8 weeks
Diastolic BP(mmHg) | 8 weeks
  Change during 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sang Yeoup Lee, MD, PhD, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, Gyeungsangnam-do, South Korea

IPD SHARING:
Plan to Share IPD: No